CLINICAL TRIAL: NCT01073514
Title: Clinical Trial of Bile Etiology,Proteomics and Metabonomics of Malignant Biliary Obstruction
Brief Title: Clinical Trial of Bile Etiology ,Proteomics and Metabonomics of Malignant Biliary Obstruction
Acronym: MBO-IR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TMU-CIH-IR-001; ChiCTR-ONC-00000752 (Registry Identifier: Chinese Clinical Trial Register(http://www.chictr.org))
Record Dates: First submitted 2010-02-21; First posted 2010-02-23 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2010-02

CONDITIONS: Malignant Biliary Obstruction
Keywords: Malignant biliary obstruction (MBO)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bile,blood and urine specimen
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To investigate bile culture and susceptibility test in patients with malignant biliary obstruction (MBO) or relation between bile, portal vein or vein culture and biliary infection. Also to get the information of bile metabonomics to find potential tumor marker .Culture of the organism is recognized as the "gold standard" for diagnosis of infection. Our research may be one of the first research on culture and susceptibility test in patients with MBO. The results of the trial research will be benefit to experiential therapy of MBO with biliary infection and diagnosis of MBO.

DETAILED DESCRIPTION:
We will obtain bile sample for culture and susceptibility ,proteomics metabonomics test after PTBD. Also get the blood and urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Those with MBO who can receive Percutaneous Transhepatic Biliary Drainage(PTBD)

Exclusion Criteria:

* Those with MBO who cannot receive Percutaneous Transhepatic Biliary Drainage(PTBD)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Malignant obstructive jaundice (MBO)
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-12; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: YU HAI PENG, MD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital; GUO ZHI, Professor, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institude and Hospital, Tianjin, Tianjin Municipality, China